CLINICAL TRIAL: NCT00301041
Title: The Relationship Between Plasma Transforming Growth Factor-beta 1 (TGF-β) and Fractionation in Radiotherapy for Breast Cancer: A Randomized Study
Brief Title: Radiation Therapy in Treating Women With Invasive Breast Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000465214
Record Dates: First submitted 2006-03-08; First posted 2006-03-10 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: Breast Cancer
Keywords: invasive ductal breast carcinoma; invasive lobular breast carcinoma; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Ductal, Breast; Carcinoma, Lobular | interventions — Chemotherapy, Adjuvant; Radiotherapy

INTERVENTIONS:
Other: laboratory biomarker analysis
Procedure: adjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Giving radiation therapy in different ways may kill more tumor cells.

PURPOSE: This randomized clinical trial is studying the side effects and best way to give radiation therapy and to see how well it works in treating patients with invasive breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the ratio between post- and pre-treatment plasma transforming growth factor-beta 1 (TGF-β) in women with invasive breast cancer undergoing hypofractionated radiotherapy vs standard-fractionated external-beam radiotherapy.

Secondary

* Establish longitudinal serum and plasma biorepository for retrospective evaluation of TGF-β and other biomarkers with special relevance to radiation response.
* Correlate pre-treatment plasma TGF-β levels with clinical fibrosis development.

OUTLINE: This is a randomized study. Patients are randomized to 1 of 2 treatment arms.

* Arm I (hypofractionated radiotherapy): Patients undergo external-beam radiotherapy once daily 5 days a week for up to 3.5 weeks (16 fractions total).
* Arm II (standard fractionated radiotherapy): Patients undergo radiotherapy as in arm I at a lower dose for up to 5 weeks (25 fractions total).

After completion of study treatment, patients are followed every 6 months for 2 years and then annually for 3 years.

PROJECTED ACCRUAL: A total of 100 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive breast cancer
* Underwent lumpectomy (breast-preserving surgery) with or without adjuvant chemotherapy within the past 12 weeks

  * Histologically negative surgical margins (i.e., no tumor on ink)
* Candidates for postoperative breast radiotherapy

  * Determined not to need radiotherapy to regional nodes (e.g., third supraclavicular field)
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of scleroderma or systemic lupus erythematosis
* No other prior or concurrent malignancy except nonmelanoma skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior breast radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-04; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine C. Park, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States